CLINICAL TRIAL: NCT04255264
Title: Adipose Tissue Inflammation and Diabetes Development (Fettvävsinflammation Och Diabetesutveckling)
Brief Title: Adipose Inflammation and Diabetes (FAB)
Acronym: FAB
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-04046
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study patients: Obese subjects scheduled to undergo abdominoplasty surgery are included. These are later classified according to metabolic status.

SUMMARY:
The study investigates whether the addition of resolution molecules can inhibit inflammation and insulin resistance in human tissue taken from obese individuals, and whether the results of these studies correlate with patient-specific resolution phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-40 kg/m2
* Ptos (i.e. excess skin) > 3 cm
* Patient underwent gastric bypass surgery >2 years ago
* Patient has had a stable weight ≥6 months at the time of operation
* Patient does not smoke (min 6 weeks prior to surgery)

Exclusion Criteria:

* Patients who do not understand spoken and written Swedish
* American Society of Anesthesiologists (ASA) classification ≥ 3
* Neurological, orthopedic or rheumatologic injury or illness affecting physical ability
* Preoperatively known hernia requiring surgical operation
* Severe mental illness

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The patients participating in this study must have undergone a gastric bypass surgery >2 years ago, and currently have excess skin of > 3 cm, thus requiring an abdominoplasty surgery. We only include patients that are obese (BMI 30-40 kg/m2). Patients interested in participating in the study donate the skin and adipose tissue that is discarded during surgery. In addition, they donate blood samples prior to surgery.
Sampling Method: Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Inflammatory status | 2025
  The inflammatory status will be studied in obese patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No